CLINICAL TRIAL: NCT01931137
Title: A Trial Investigating the Pharmacokinetics and Pharmacodynamics of NNC0123-0000-0338 in a Tablet Formulation With Three Different Coatings in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1953-3973; 2012-004202-10 (EudraCT Number); U1111-1134-6321 (Other: WHO)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Coating A (Experimental): Each subject will in random order be allocated to three single-dose administrations of insulin 338 in a GIPET® I tablet with 3 different coatings, respectively, on three separate dosing visits (Visits 2, 3 and 4). Each of the three dosing days will be separated by a 3-week wash-out period (ranging from 20 to 28 days)
  Interventions: Drug: insulin 338 (GIPET I)
- Coating B (Experimental): Each subject will in random order be allocated to three single-dose administrations of insulin 338 in a GIPET® I tablet with 3 different coatings, respectively, on three separate dosing visits (Visits 2, 3 and 4). Each of the three dosing days will be separated by a 3-week wash-out period (ranging from 20 to 28 days)
  Interventions: Drug: insulin 338 (GIPET I)
- Coating C (Experimental): Each subject will in random order be allocated to three single-dose administrations of insulin 338 in a GIPET® I tablet with 3 different coatings, respectively, on three separate dosing visits (Visits 2, 3 and 4). Each of the three dosing days will be separated by a 3-week wash-out period (ranging from 20 to 28 days)
  Interventions: Drug: insulin 338 (GIPET I)

INTERVENTIONS:
Drug: insulin 338 (GIPET I) — Dose level of 8100 nmol will be orally administered as one tablet per dose.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of NNC0123-0000-0338 (insulin 338) in a tablet formulation with three different coatings in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0-28.0 kg/m^2 (both inclusive)
* Subject who is considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, ECG (electrocardiogram) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as informed consent
* Presence of clinically significant acute gastro-intestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to first dosing, as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin 338 concentration-time curve | From dosing to infinity calculated from a 0-288 hours NNC0123-0000-0338 serum concentration-time-curve based on 38 sampling time points.

SECONDARY OUTCOMES:
Area under the serum insulin 338 concentration-time curve | From 0 to 288 hours after a single dose (SD)
Area under the glucose infusion rate (GIR)-time curve | From 0 to 24 hours after a single dose
Number of treatment emergent adverse events | As recorded from trial product administration (Day 1) at Sub-visit A and until Sub-visit G (Day 13)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com